CLINICAL TRIAL: NCT06612723
Title: High vs Low-frequency of High-intensity Training in Chronic Stroke
Acronym: F-ITT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Responsible Party: Principal Investigator, George Hornby, Professor, Indiana University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 24114
Record Dates: First submitted 2024-09-20; First posted 2024-09-25 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Stroke
Keywords: stroke; gait; rehabilitation; high-intensity; frequency
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High frequency (Experimental): Individuals will receive up to 18 visits of high-intensity gait training and activity coaching over 6 weeks
  Interventions: Other: high-intensity gait training; Behavioral: Physical activity coaching
- Low frequency (Active Comparator): Individuals will receive up to 18 visits of high-intensity gait training and activity coaching over 12 weeks
  Interventions: Other: high-intensity gait training; Behavioral: Physical activity coaching

INTERVENTIONS:
Other: high-intensity gait training — Individuals will perform up to 40 minutes of walking practice during 60 minute sessions while targeting heart rates of at least 70% heart rate reserve.
Behavioral: Physical activity coaching — Individuals will receive feedback on the minutes of walking activity performed on non-training days and provided coaching strategies to increase this metric.

SUMMARY:
The purpose of this pilot study is to investigate the potential role of training frequency on locomotor outcomes following high-intensity gait training and provision of a home walking program.

DETAILED DESCRIPTION:
This study will utilize a 2 arm randomized trial to investigate potential differences in locomotor and community outcomes following 18 visits of high-intensity gait training provided over 6 weeks (high frequency) or 12 weeks (low frequency). Following confirmation of eligibility and baseline testing, individuals will be randomized to either high or low frequency of training and complete subsequent testing at 6 weeks, 12 weeks, and 24 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Unilateral deficits following stroke > 6 months prior; however individuals > 4 months post-stroke are eligible for consenting, but final eligibility and potential enrollment will not occur until > 6 months
* Age 18-85
* Weight < 350 pounds
* Able to follow 3-step commands
* Able to ambulate with self-selected gait speeds between 0.10-1.0 m/s without physical assistance, but with below knee bracing and/or assistive device as needed
* Lower extremity Fugl-Meyer < 34
* Medical clearance to participate

Exclusion Criteria:

* Evidence of cerebellar ataxia
* Uncontrolled cardiopulmonary or metabolic disease that limits exercise participation, active heterotopic ossification, recurrent history of lower extremity fractures, previous orthopedic or other peripheral or central neurologic injury that may impair locomotor activities such that, in the judgement of the PI, could compromise the safety of the participant, limit the ability to complete the study, or compromise the objectives of the study.
* Currently participating in other physical therapy
* >50 units of Botox in the lower extremity OR in the lower extremity, but above the knee if the participant wears an ankle-foot-orthosis (AFO) within the past three months

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-09-16 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
6-minute walk test | After 12 weeks
  Individuals will be asked to "cover as much ground as possible" over 6 mins. Heart rate will additionally be measured during this assessment (distance in m)

SECONDARY OUTCOMES:
Peak treadmill speed | After 12 weeks
  Individuals will participate in a walking-based graded exercise test. While harnessed for safety, a motorized treadmill will be initially set to 0.1 m/s and increased by 0.1 m/s each minute until the test is terminated due: 1) requests to stop, 2) unable to keep up with the treadmill and/or loses their balance, 3) absolute exercise test termination criteria provided by ACSM. The highest speed that the individual can walk for a minute at is the peak treadmill speed.

OTHER OUTCOMES:
Functional Gait Assessment | After 12 weeks
  10 item assessment of dynamic balance. Example tasks include walking with head turns, with eyes closed, and walking backwards.
30 second Sit to Stand Test | After 12 weeks
  Participants will be asked to rise from a chair without using their arms and then return to sitting as many times as possible in 30 seconds.
Activity-Specific Balance Confidence (ABC) Scale | After 12 weeks
  This questionnaire asks individuals to rate their balance-confidence from 0 (no confidence) to 100 (completely confident) during a variety of 16 commonly performed tasks such as walking around a house or getting into a car.
Oxygen Consumption | After 12 weeks
  Oxygen consumption will be measured via a portable metabolic cart (K5; COSMED) during the previously described graded exercise test. Participant will wear a snug fitting mask that covers their mouth and nose, but does not affect the amount or quality of air that they breathe. The mask will be connected to a small backpack that collects information on the rate of breathing and oxygen consumed.
Medical Outcomes Survey Short-Form 36 (SF-36) | After 12 weeks
  This 36-question survey asks individuals about how their current health may limit their ability to perform typical physical and social activities.
Steps per Day | After 12 weeks
  Participants will wear a research-grade pedometer (StepWatch; Modus Health) during waking hours for ~1-2 weeks before beginning the training protocol, during the intervention period, and after completing training protocol to quantify home and community mobility. Participants will also be asked to document their daily minutes walked for exercise, number of walking bouts, where they performed the activity, and subjectively how hard they were working while walking for exercise.
Gait speed | After 12 weeks
  This is an assessment of overground walking speed measured across a distance of ~20 feet and will be conducted at both self-selected (instructions: "walk at your usual, comfortable pace") and fastest (instructions: "walk as fast as you safely can") walking speeds on a pressure sensitive mat (speed in m/s; Zeno Walkway).

CONTACTS AND LOCATIONS:
Overall Officials: Thomas G Hornby, PhD, Principal Investigator — Indiana University
Locations (1):
- Rehabilitation Hospital of Indiana, Indianapolis, Indiana, United States